CLINICAL TRIAL: NCT04149353
Title: Utility of PET/MR in Surgical Planning for Breast Cancer Treated With Neoadjuvant Chemotherapy
Brief Title: PET/MR in Surgical Planning for Breast CA Treated With Neoadj Chemo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1716
Record Dates: First submitted 2019-03-14; First posted 2019-11-04 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PET/MR (Experimental): Each patient will undergo two combined PET/MR scans. The pre-treatment and post-treatment combined PET/MR scans are for research purposes and not part of the patient's standard of care.
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — Patient will be scheduled for a pre-treatment PET/MR and proceed to neoadjuvant chemotherapy per the direction of the medical oncologist. Within four weeks after completion of chemotherapy the patient will undergo a post-treatment PET/MR, and proceed for curative intent surgery if they are still surgical candidates.

SUMMARY:
Purpose: To assess the utility of combined, simultaneous positron emission tomography (PET) and magnetic resonance imaging (MRI), collectively called PET-MR, in assessing response to neoadjuvant chemotherapy and surgical treatment decisions for operable breast cancers.

Participants: Adult patients with operable breast cancer that are being treated at UNC with neoadjuvant chemotherapy followed by potentially curative surgical resection.

Procedures (methods): Patients who are being treated with neoadjuvant chemotherapy followed by surgical resection and for whom pre- and post-treatment MR imaging is part of planned treatment will undergo additional pre-treatment and post-treatment PET/MR. The response to treatment will be assessed at post-treatment by evaluating change in tumor size from MRI, change in response to dynamic contrast enhanced (DCE) MRI, and 18F-fluorodeoxyglucose (18F-FDG) avidity from PET. Patients will then undergo surgery. Their pathology will be reviewed for treatment effect as assessed by residual cancer burden (RCB) score. Patients will be followed and assessed for recurrence.

DETAILED DESCRIPTION:
Investigators propose that the changes indicated by PET/MR imaging from pre-treatment to post-treatment time points will accurately predict the patient's response to neoadjuvant chemotherapy, providing useful prognostic and surgical-planning information. The study will enroll patients with operable breast cancer being treated with neoadjuvant chemotherapy followed by potentially curative surgical resection. The standard of care for these patients would not normally include PET imaging but may include MR imaging. Patients in the study will receive combined PET/MR imaging prior to treatment and following treatment. Then, patients will receive curative intent surgery and be followed in the usual fashion and assessed for local and/or distant recurrent disease. The pathology report will be reviewed for therapy treatment effect as assessed by Residual Cancer Burden (RCB) score. Quantitative measures from PET and MRI will be computed: the change in PET tumor-mean standardized uptake value (SUV) and tumor size as assessed by MRI, from pre- to post-treatment. The image-based quantitative measures will be correlated with the pathology outcomes to evaluate predictability of the image measures for RCB score. Patients will be followed with the intent of further correlating image measures with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age (no upper age limit)
* Signed, IRB-approved written informed consent
* Must have clinical T1-3, N0-3, M0 disease. All phenotypes are acceptable..
* Must have surgically curable disease as evaluated by the UNC Multidisciplinary Tumor Board.
* Must have pre- and post-treatment MRI imaging as part of the treatment plan.
* Must be able to meet size restrictions for the PET-MR scanner: chest depth and abdominal depth less than 27 cm (approximately the smallest 55% of women will meet this), as measured on imaging or with physical template.
* Must be in acceptable health to undergo chemotherapy and curative intent surgery as assessed by Multidisciplinary Tumor Board.
* Must be able to understand and comply with study procedures for the entire length of the study.
* Must receive their chemotherapy and curative intent surgery at UNC Hospitals. -If patient has a history of prior malignancy, including melanoma, patient must be cancer- free for three or more years. Non-melanoma skin cancers will be included even if not cancer-free for three years.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to each PET/MRI

Exclusion Criteria:

* Inability to tolerate MRI (e.g., inability to lie flat for >1 hour)
* Presence of pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes or near pelvis that would create excessive imaging artifact
* Poorly controlled diabetes mellitus
* Patient receiving neoadjuvant endocrine therapy (due to low likelihood of complete response)
* Pregnancy or lactating female
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study
* Evidence of distant disease on physical exam or initial imaging
* Medical conditions precluding chemotherapy or curative intent surgery
* Incarcerated or otherwise institutionalized at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lalush, PhD, Principal Investigator — UNC Biomedical Engineering
Locations (1):
- UNC- Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Cancer Patients: Patients who are being treated with neoadjuvant chemotherapy followed by surgical resection and for whom pre- and post-treatment MR imaging is part of planned treatment.
Period: Overall Study
Arm/Group | Breast Cancer Patients
Started | 1 (The study was terminated for low recruitment before this subject's second imaging scan was due.)
Completed | 0
Not Completed | 1
Not completed — Study terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1
Pre-surgery PET-MR scan tumor size [Mean (Standard Deviation); unit: millimeters] | 4 (0)

OUTCOME MEASURES:

1. Primary Outcome: Change in PET Activity Estimates From Pre-treatment to Post-treatment
Description: Primary endpoint is the determination of the potential for PET activity estimates to predict RCB score in comparison with that of dynamic contrast enhanced (DCE) MRI. Treatment response will be determined on final pathological evaluation of the resected specimens by way of the RCB score.
Time Frame: Time Frame: Changes in image measures will be assessed from baseline scans, prior to therapy, to post-treatment scans, taken six months after baseline. Pathology data will be obtained post-surgery.
Population: Single subject did not complete the second scan, so outcome measure could not be assessed.
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Performance of Metrics Combining Multiple Features From PET and MR in Prediction of Response to Therapy
Description: Quantitative image measures from PET and MR will be compiled and an optimal linear regression will be derived between the image metrics and the outcome measure from pathology, the RCB score. Prediction performance of the regression relation will be assessed using a leave-one-out cross-validation approach.
Time Frame: Changes in image measures will be assessed from baseline scans, prior to therapy, to post-treatment scans, taken six months after baseline. Pathology data will be obtained post-surgery.
Population: Single subject did not complete the second scan, so outcome measure could not be assessed.
Groups:
- Breast Cancer Patients: Each patient will undergo two combined PET/MR scans. The pre-treatment and post-treatment combined PET/MR scans are for research purposes and not part of the patient's standard of care.
  PET/MR: Patient will be scheduled for a pre-treatment PET/MR and proceed to neoadjuvant chemotherapy per the direction of the medical oncologist. Within four weeks after completion of chemotherapy the patient will undergo a post-treatment PET/MR, and proceed for curative intent surgery if they are still surgical candidates.
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Breast Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04149353/Prot_SAP_000.pdf